CLINICAL TRIAL: NCT01691222
Title: Percutaneous Tracheostomy in Intensive Care Unit With a Dedicated Double Lumen Endotracheal Tube
Brief Title: Tracheostomy in ICU With a Double Lumen Endotracheal Tube
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, Paolo Pelosi, Full Professor chair of Anesthesiology and Intensive Care Medicine. Chief of Intensive Care Unit, University of Genova
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 90/12
Record Dates: First submitted 2012-08-30; First posted 2012-09-24 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Acute Respiratory Failure; Heart Failure; Neurological Disease
Keywords: Bedside percutaneous tracheostomy; Intensive Care Unit; Dedicated Double-lumen tube; Ineffective Airway Clearance; weaning failure
MeSH Terms: conditions — Heart Failure; Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Double lumen endotracheal tube tracheostomy (Other): Tracheostomy with a dedicated double lumen endotracheal tube
  Interventions: Device: Double lumen endotracheal tube tracheostomy

INTERVENTIONS:
Device: Double lumen endotracheal tube tracheostomy — Percutaneous tracheostomy in this study will be performed with the use of a dedicated double-lumen endotracheal tube.
  The dedicated double-lumen endotracheal tube (Deas S.R.L, Italy) has an upper and a lower lumen. The upper one will be occupied by flexible fiberoptic bronchoscope while the lower one is exclusively dedicated to patient ventilation during the procedure. The lower lumen has a a semi-elliptical cross section. This tube will be placed in the patient airway with a direct laryngoscopy. After this intubation, a percutaneous dilatational tracheostomy will be performed with the standard techniques recognised in the literature.
  Other Names: International Patent n° PCT/IT2012/000154

SUMMARY:
Percutaneous tracheostomy in Intensive care unit (ICU) is performed with the use of flexible fiberoptic bronchoscope inside the conventional single lumen endotracheal tube owned by the patients. This situation may lead to many disadvantages for ventilation and airway protection of critically ill patients during the procedures. The use of double lumen endotracheal tube dedicated to the percutaneous tracheostomies may:

1. improve the ventilation of patients during the procedure,
2. protect the posterior tracheal wall from damage related to the different step of tracheostomies,
3. protect the lungs from blood and secretions coming down from the chosen site of tracheostomy.

So the aim of this study is to evaluate the oxygenation, gas exchange, ventilation and complications of percutaneous tracheostomies performed in ICU with a dedicated double lumen endotracheal tube.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years and at least one of following criteria:
* prolonged endotracheal intubation
* prolonged mechanical ventilation
* difficult/prolonged weaning
* inability to protect the airway

Exclusion Criteria:

* infection of neck tissues
* previous surgical neck interventions
* recent surgical interventions or fracture of the cervical spine

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
change in gas-exchange | at the baseline and the end of the procedure (average time expected for the procedure is 30 minutes)
  The investigator will perform an arterial blood gas to evaluate PaO2/FiO2 ratio

SECONDARY OUTCOMES:
change in arterial carbon dioxide | at the baseline and at the end of the procedure (average time expected for the procedure is 30 minutes)
  the investigator will perform an arterial blood gas to evaluate PaCO2
change in peak airway pressure | at the baseline and at the end of the procedure (average time expected for the procedure is 30 minutes)
  the investigator will record peak airway pressure
change in plateau airway pressure | at the baseline and at the end of the procedure (average time expected for the procedure is 30 minutes)
  the investigator will record plateau airway pressure
change in air-trapping | at the baseline and at the end of the procedure (average time expected for the procedure is 30 minutes)
  the investigator will record auto-PEEP at the of expiration as a measure of air-trapping
early complications | in the first 24 hours from the end of the procedure
  early complications are:multiple intubation attempts (more than 1), accidental extubation, paratracheal insertion, injuries to blood vessels in the neck, oesophageal injury, accidental decannulation, malposition of the tracheostomy tube, tracheal cuff puncture, multiple punctures (more than 1), surgical conversion and percutaneous tracheostomy failure, minor bleeding (compressible), major bleeding (incompressible), pneumothorax,
late complications | from the 2nd day ofter the procedure until the ICU discharge (expected average of 2 weeks)
  late complications are: minor bleeding (compressible), major bleeding (incompressible) tracheostomy puncture site infection, subglottic stenosis, fracture of a tracheal cartilage, granuloma.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pelosi, Professor, Study Director — Universita degli Studi di Genova; Giuseppe Servillo, Professor, Study Director — Federico II University
Locations (2):
- Italy (2):
  - University of Genoa, Genoa, Italy
  - University of Naples "Federico II", Naples, Italy

REFERENCES:
- [Background] Rana S, Pendem S, Pogodzinski MS, Hubmayr RD, Gajic O. Tracheostomy in critically ill patients. Mayo Clin Proc. 2005 Dec;80(12):1632-8. doi: 10.4065/80.12.1632. PMID 16342657
- [Background] De Leyn P, Bedert L, Delcroix M, Depuydt P, Lauwers G, Sokolov Y, Van Meerhaeghe A, Van Schil P; Belgian Association of Pneumology and Belgian Association of Cardiothoracic Surgery. Tracheotomy: clinical review and guidelines. Eur J Cardiothorac Surg. 2007 Sep;32(3):412-21. doi: 10.1016/j.ejcts.2007.05.018. Epub 2007 Jun 27. PMID 17588767
- [Background] King C, Moores LK. Controversies in mechanical ventilation: when should a tracheotomy be placed? Clin Chest Med. 2008 Jun;29(2):253-63, vi. doi: 10.1016/j.ccm.2008.01.002. PMID 18440435
- [Background] Durbin CG Jr. Tracheostomy: why, when, and how? Respir Care. 2010 Aug;55(8):1056-68. PMID 20667153
- [Background] Mallick A, Bodenham AR. Tracheostomy in critically ill patients. Eur J Anaesthesiol. 2010 Aug;27(8):676-82. doi: 10.1097/EJA.0b013e32833b1ba0. PMID 20523214
- [Background] Ciaglia P, Firsching R, Syniec C. Elective percutaneous dilatational tracheostomy. A new simple bedside procedure; preliminary report. Chest. 1985 Jun;87(6):715-9. doi: 10.1378/chest.87.6.715. PMID 3996056
- [Background] Fantoni A, Ripamonti D. A non-derivative, non-surgical tracheostomy: the translaryngeal method. Intensive Care Med. 1997 Apr;23(4):386-92. doi: 10.1007/s001340050345. PMID 9142576
- [Background] Griggs WM, Worthley LI, Gilligan JE, Thomas PD, Myburg JA. A simple percutaneous tracheostomy technique. Surg Gynecol Obstet. 1990 Jun;170(6):543-5. PMID 2343371
- [Background] Trottier SJ, Hazard PB, Sakabu SA, Levine JH, Troop BR, Thompson JA, McNary R. Posterior tracheal wall perforation during percutaneous dilational tracheostomy: an investigation into its mechanism and prevention. Chest. 1999 May;115(5):1383-9. doi: 10.1378/chest.115.5.1383. PMID 10334157
- [Background] Campos JH. Update on tracheobronchial anatomy and flexible fiberoptic bronchoscopy in thoracic anesthesia. Curr Opin Anaesthesiol. 2009 Feb;22(1):4-10. doi: 10.1097/ACO.0b013e32831a43ab. PMID 19295287
- [Derived] Vargas M, Pelosi P, Tessitore G, Aloj F, Brunetti I, Arditi E, Salami D, Kacmarek RM, Servillo G. Percutaneous dilatational tracheostomy with a double-lumen endotracheal tube: a comparison of feasibility, gas exchange, and airway pressures. Chest. 2015 May;147(5):1267-1274. doi: 10.1378/chest.14-1465. PMID 25375865